CLINICAL TRIAL: NCT01378195
Title: iCare Stress Management e-Training for Dementia Family Caregivers
Acronym: iCare
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photozig, Inc. (Industry)
Collaborators: Stanford University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pz-A103a; R44AG032762 (NIH)
Record Dates: First submitted 2011-06-17; First posted 2011-06-22 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's Disease; Dementia; caregiving; caregiver; coping; coping with caregiving; stress
MeSH Terms: conditions — Alzheimer Disease; Dementia

ARMS (2):
- CBT-based (Experimental): CBT-based program (Cognitive Behavioral Therapy) with video, workbook, and website
  Interventions: Behavioral: CBT-based program for dementia caregivers
- Educational/Resources Materials (Active Comparator): Educational/Resources Materials: video, workbook, and website.
  Interventions: Behavioral: Educational/Resources program

INTERVENTIONS:
Behavioral: CBT-based program for dementia caregivers — Participants will receive a CBT-based program [Cognitive Behavioral Therapy], containing videos, workbook, and website.
  Arms: CBT-based
Behavioral: Educational/Resources program — Participants will receive a traditional educational/resources program, containing videos, workbook, and website.
  Arms: Educational/Resources Materials

SUMMARY:
Photozig and Stanford University are creating a program to help cope with caregiving, alleviate related stress, and enhance quality of life for caregivers, with funding from the National Institute on Aging. This home-based program includes a free DVD, printed materials, and resource website. In addition, after completing the program, participants will have free access to final online resources for 1 year. There are no face-to-face meetings, and participants can live anywhere in the United States.

DETAILED DESCRIPTION:
The goal of this study is to develop the iCare Program, a DVD/online video training that builds skills and stimulates practice. We are evaluating different materials, which may encourage caregiver participation, enable user interaction, and promote better assimilation of concepts. We are designing the program to help to enhance caregivers' skills to deal with demanding tasks of caregiving, alleviate related stress, and improve quality of life.

Research Program Steps:

1. Caregivers will be asked some simple questions about themselves and their family members to see if they are eligible for the project (fill out Enrollment Form and Informed Consent).
2. A Program survey will be sent, which can be completed online, or returned in a pre-mailed envelope.
3. A DVD, materials, link to our website, login information, and instructions will be mailed to participants. We ask participants to watch the DVD, read printed materials, use the website, and follow instructions. Materials are expected to help participants in their caregiver role.
4. After completing the program, the second and final survey should be filled out online or returned by pre-mailed envelope.

ELIGIBILITY:
Inclusion Criteria:

* Care for an individual with Alzheimer's Disease or other dementia.
* Own a DVD player or have Internet access.
* Minimum age of 21 years old.
* Spend at least 8 hours/week caring for a person with dementia, which may include assisting, watching, monitoring, or being available to help (e.g. during sleep time).

Exclusion Criteria:

* Severe psychological or physical illness.
* Inability to read and follow English instructions.
* High level of depressive symptoms.
* Unwillingness to participate in all aspects of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Kajiyama, MS, Principal Investigator — Photozig, Inc.
Locations (1):
- Photozig, Inc., Moffett Field, California, United States

REFERENCES:
- See also: Dementia Caregiving Program — http://www.icarefamily.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: May 2011 to March 2012
Pre-assignment Details: Participant assignment to group was random.
Period: Overall Study
Arm/Group | CBT-based | Educational/Resources Materials
Started | 75 | 75
Completed | 46 | 57
Not Completed | 29 | 18
Not completed — Lost to Follow-up | 29 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-based | Educational/Resources Materials | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 48 | 95
  >=65 years | 28 | 27 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 66 | 125
  Male | 16 | 9 | 25
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Perceived Stress Scale
Description: The "Perceived Stress Scale" measures the overall level of stress. This instrument contains 10 items accessing overall appraisals of stress in the past month. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=40. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-based | Educational/Resources Materials
Number analyzed (Participants) | 46 | 57
units on a scale | 15.83 (5.07) | 16.41 (7.15)

2. Secondary Outcome: Revised Memory and Behavior Problems Checklist
Description: This scale measures the type/number of dementia patients disturbing behaviors, and how much they bother caregivers with 24 items describing possible troublesome behaviors that the patient might evidence in the past month. Caregivers are first asked whether the dementia patient had displayed any of these in the time period, and secondly to rate on a 5-point scale (0=not at all; 4= extremely) how much this "bothered or upset" them. A "conditional bother" score is calculated which is the "upset" or "bother" ratings for only the problematic behavior that occurred. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=4. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-based | Educational/Resources Materials
Number analyzed (Participants) | 46 | 57
units on a scale | 0.83 (0.63) | 0.91 (0.75)

3. Secondary Outcome: Perceived Quality of Life
Description: The "Perceived Quality of Life" (PQoL instrument) measures quality of life by the evaluation of major categories of fundamental life needs. This measure was developed using a normative sample of older individuals, and has been used in a number of studies investigating the effects of chronic disorders on the perceived quality of life. The scale contains items describing level of satisfaction with needs and resources in various categories. The scale refers to the caregiver. Minimum (worst value) = 0. Maximum score (best value=10. Higher values represent a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-based | Educational/Resources Materials
Number analyzed (Participants) | 46 | 57
units on a scale | 6.34 (1.54) | 6.31 (1.84)

ADVERSE EVENTS:
Arm/Group | CBT-based | Educational/Resources Materials
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes